CLINICAL TRIAL: NCT02955511
Title: Comparison of 3 Direct Laryngoscopes: Inscope DL Blade Size 3.5 and DL Blade 3.5 Sun-Med GreenLine®/D™ to DL Blade 3 Sun-Med GreenLine®/D™ for Tracheal Intubation in Patients Undergoing Lumbar Spine Surgery, a Prospective Randomized Study
Brief Title: Comparison of 3 Direct Laryngoscopes for Tracheal Intubation in Patients Undergoing Lumbar Spine Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The blade used in the study was modified (changed) by the manufacturer, it does not longer exist.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Professor, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: Pro00045198
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Anesthesia; Airway

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Blade MAC size 3 (Active Comparator): Patient will be intubated using a:
  Direct Laryngoscope (DL) Mac size 3 (Sun-Med GreenLine®/D™ Macintosh)
  Interventions: Device: Blade MAC size 3
- Blade MAC size 3.5 (Active Comparator): Patient will be intubated using a:
  DL-blade mac size 3.5 (Sun-Med Greenline®/D™ Macintosh)
  Interventions: Device: Blade MAC size 3.5
- Inscope Blade size 3.5 (Experimental): Patient will be intubated using a:
  Inscope DL-blade size 3.5
  Interventions: Device: Inscope Blade size 3.5

INTERVENTIONS:
Device: Blade MAC size 3 — Patient will be intubated using the DL- Blade MAC size 3
  Arms: Blade MAC size 3
Device: Blade MAC size 3.5 — Patient will be intubated using the DL- Blade MAC size 3.5
  Arms: Blade MAC size 3.5
Device: Inscope Blade size 3.5 — Patient will be intubated using the Inscope Blade size 3.5
  Arms: Inscope Blade size 3.5

SUMMARY:
Hypothesis The use of Macintosh blade sized #3.5 (vs Macintosh size #3) would reduce the time required to achieve successful tracheal intubation and improve the glottic view.

Study objective The purpose of this research study is to compare 3 different laryngoscope blades (sizes: 3.5, 3.5 and 3) and see if the blades size 3.5 will reduce the time required to achieve successful tracheal intubation and improve the physician's view of the glottis compared to the standard direct laryngoscope using the blade size 3, in patients undergoing lumbar surgery.

Primary end point: time to achieve successful tracheal intubation.

Secondary end points: glottic view at intubation, number of intubation attempts and effectiveness of the integrated suction in the Inscope Direct Laryngoscope.

DETAILED DESCRIPTION:
Laryngoscopy is a common medical procedure used during elective and emergency intubations. The procedure is performed with either a direct or video laryngoscope with the device selected dependent on tool availability, provider (i.e. anesthesiologist, emergency physician, ENT physician, paramedic, etc.) preference, patient characteristics, and intubation difficulty. The direct laryngoscope technique involves a line-of-sight view from the patient's mouth to vocal cords along the blade of the scope. The direct laryngoscopy technique is the oldest technique associated with intubation. However, despite continuous improvements to direct laryngoscope size and shape since its inception in the late 19th century, no improvement yet addresses one major problem with airway visualization: the provider will experience a difficult intubation if liquids (i.e. gastric content, blood, mucus, etc.) obstruct the view.

The Sun-Med GreenLine®/D™ Macintosh is a line of disposable direct Macintosh laryngoscopes. It features a stainless steel blade and polycarbonate light-pipe to direct light into the airway. The handle, with integrated batteries and LED light, and blade are separately packaged prior to use. The GreenLine®/D™ Macintosh line is available in the standard sizes (0, 1, 2, 3, 4) and a new size built to improve blade sizing for many adults 3.5 when a Mac 3 is too short, but a Mac 4 is too large. The GreenLine®/D™ Macintosh does not feature integrated suction.

The Inscope Direct Laryngoscope (developed by Inscope Medical Solutions) is a new disposable direct laryngoscope with two integrated and controllable (flow on/off) suction pathways. By integrating controllable suction with two independent pathways into the laryngoscope, the provider is able to select the primary (blade tip) suction pathway to clear secretions ahead of the laryngoscope and the secondary (at blade mid-length, below blade) to prevent and clear fluids that may re-accumulate during the procedure. Integrating the suction into the device prevents the common current practice of "juggling" the current suction catheter and endotracheal (breathing) tube in one hand while holding the patient's airway open with the other hand. While the incidence of aspiration of fluids into the lungs as a result of poor airway fluid management is low, the outcomes associated with this complication are very poor.

The Inscope Direct Laryngoscope has been developed as a Macintosh 3.5 sized blade to meet the size requirements of the majority of patients. This assumption is backed up by a trend among disposable direct laryngoscope manufacturers toward the 3.5 blade size, with at least 5 creating a 3.5 blade, including Teleflex, Sun-Med, Flexicare, Mercury Medical, and Curaplex.

This study will compare the Inscope Direct Laryngoscope (blade size 3.5) with the currently used standard single-use Sun-Med Greenline/D Macintosh laryngoscopes DL-blade mac size and Sun-Med Greenline/D-blade size 3.5.

All Direct Laryngoscopes are considered a Class I exempt device by the FDA. Because the risks associated with laryngoscopes are well known and documented, they are considered a non-significant risk device for studies involving humans.

ELIGIBILITY:
A. Inclusion Criteria:

1. Patients undergoing lumbar spine surgery procedures under general anesthesia
2. Patients with a documented BMI of <35
3. Willingness and ability to sign an informed consent document
4. 18 - 80 years of age of either gender
5. American Society of Anesthesiologists (ASA) physical status classification I - II or III

B. Exclusion Criteria:

1. Patients who are deemed to be such a significant of an airway risk that they necessitate awake fiberoptic intubation or a difficult tracheal intubation is anticipated
2. Patients with history of difficult intubation
3. Patients with oxygen saturation less than 95% at room air
4. Patients with history facial abnormalities, oral-pharyngeal cancer or reconstructive surgery
5. Any pathologies of the mouth, pharynx or larynx, or the access to the airway is restricted
6. Patients with Immobilized cervical spine, or history of cervical abnormalities
7. Patients with a history of uncontrolled gastroesophageal reflux, hiatus hernia or diabetic gastroparesis
8. Any coagulation disorder
9. Pregnant patients
10. Emergency surgeries
11. Any other conditions or use of any medication which may interfere with the conduct of the Study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Blade MAC Size 3: Patient will be intubated using a:
  Direct Laryngoscope (DL) Mac size 3 (Sun-Med GreenLine®/D™ Macintosh)
  Blade MAC size 3: Patient will be intubated using the DL- Blade MAC size 3
- Blade MAC Size 3.5: Patient will be intubated using a:
  DL-blade mac size 3.5 (Sun-Med Greenline®/D™ Macintosh)
  Blade MAC size 3.5: Patient will be intubated using the DL- Blade MAC size 3.5
- Inscope Blade Size 3.5: Patient will be intubated using a:
  Inscope DL-blade size 3.5
  Inscope Blade size 3.5: Patient will be intubated using the Inscope Blade size 3.5
Period: Overall Study
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
Started | 1 | 3 | 1
Completed | 1 | 3 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5 | Total
Number analyzed (Participants) | 1 | 3 | 1 | 5
Age, Customized [Count of Participants; unit: Participants]
  50 to 64 years | 1 | 1 | 0 | 2
  65 to < 75 years | 0 | 1 | 0 | 1
  >= 75 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — The study terminated early and did not have sufficient enrollment (only five total) into an arm of the study to produce any meaningful results.
  Participants
    Female | 0 | 1 | 1 | 2
    Male | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Description: The study terminated early and did not have sufficient enrollment (only five total) into an arm of the study to produce any meaningful results.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 3 | 1 | 4
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time (Using a Stopwatch)
Description: Intubation Time:
  It is the time taken to intubate: from the initial insertion of the laryngoscope blade to the placement of the tracheal tube (approximately 3 minutes).
  An intubation attempt:
  It is defined as the insertion of the laryngoscope blade into a patient's mouth, with the objective of inserting an endotracheal tube into the trachea.
Time Frame: up to 3 minutes
Population: Measure Description:
  The study was terminated early, only FIVE (5) subjects total were enrolled for the three arms groups. It is impossible to produce meaningful results having only five subjects enrolled.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
Number analyzed (Participants) | 1 | 3 | 1
Seconds | 38 (0) | 15.3 (2) | 17 (0)

2. Primary Outcome: Glottis Visualization POGO Score
Description: The percentage of the glottis visualized (POGO) score It represents the percentage of glottic opening seen; the score ranges from 0% when none of the glottis is seen to 100% when the entire glottis, including the anterior commissure, is seen.
Time Frame: During intubation procedure, up to 1 minute
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of glottic opening
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
Number analyzed (Participants) | 1 | 3 | 1
percentage of glottic opening | 75 (0) | 96.6 (4) | 80 (0)

3. Primary Outcome: Time From the Insertion of the Laryngoscope Blade to Confirm w/ CO2 Waveform
Description: The time following the initial insertion of the laryngoscope blade into the mouth to confirm w/ CO2 waveform
Time Frame: During intubation procedure, up to 3 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
Number analyzed (Participants) | 1 | 3 | 1
Seconds | 49 (0) | 36.5 (12) | 26 (0)

4. Secondary Outcome: Intubation Attempts
Description: An intubation attempt is defined as the insertion of the laryngoscope blade into a patient's mouth, with the objective of inserting an endotracheal tube into the trachea.
  The number of intubation attempts in each participant for successful tracheal intubation measured how many times the anesthesiologist attempted to place the tube into the trachea of each patient.
Time Frame: 3 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Intubation Attempts
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
Number analyzed (Participants) | 1 | 3 | 1
Intubation Attempts | 1 (0) | 1 (0) | 1 (0)

5. Secondary Outcome: Glottis Visualization Using Cormack Lehane
Description: Grade Description Approximate frequency Likelihood of difficult intubation
  1. Full view of glottis 68-74% <1%
  2. a Partial view of glottis 21-24% 4.3-13.4%
  2b Only posterior extremity of glottis seen or only arytenoid cartilages 3.3-6.5% 65-67.4% 3 Only epiglottis seen, none of glottis seen 1.2-1.6% 80-87.5% 4 Neither glottis nor epiglottis seen very rare
  Note:
  In the analysis of the data collected for 5 participants, there was no differentiation between "2a" and "2b" for a grade of "2."
Time Frame: During intubation procedure, up to 1 minute
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
Number analyzed (Participants) | 1 | 3 | 1
score on a scale | 2 (0) | 1.3 (0.6) | 2 (0)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Blade MAC Size 3 | Blade MAC Size 3.5 | Inscope Blade Size 3.5
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT02955511/Prot_003.pdf
  • Statistical Analysis Plan (2016-11-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT02955511/SAP_004.pdf